CLINICAL TRIAL: NCT06030570
Title: PROGRESS: The Effect of an Interdisciplinary Program for Rehabilitation for Spinal Disorders
Brief Title: Effect of an Interdisciplinary Spine Rehabilitation Program
Acronym: PROGRESS
Status: Recruiting | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Sofie Rummens, Principal Investigator, Physical and Rehabilitation Medicine Specialist, PhD in Biomedical Sciences, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S67679
Record Dates: First submitted 2023-08-24; First posted 2023-09-11 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Low Back Pain; Spine Disease
MeSH Terms: conditions — Low Back Pain; Spinal Diseases | interventions — Rehabilitation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with low back pain: Patients of University Hospitals Leuven participating in the interdisciplinary spine rehabilitation program (REVITA)
  Interventions: Other: Rehabilitation program (Revita)

INTERVENTIONS:
Other: Rehabilitation program (Revita) — Multidisciplinary programs in an outpatient hospital setting are coordinated by specialists in Physical and Rehabilitation Medicine. These programs combine a physical part (e.g., specific exercises, manual techniques) with at least one other element (psychological, social, educational or occupational intervention). In a multidisciplinary spine rehabilitation program, a maximum of 36 sessions over a maximum time period of 6 months is offered. Afterwards, a (monodisciplinary) follow-up trajectory (K15) is possible, consisting of maximum 104 sessions a year.

SUMMARY:
The goal of this research project is to evaluate the effectiveness of the current interdisciplinary rehabilitation program (Revita) and follow-up trajectory for chronic lumbar spine disorders in the University Hospitals Leuven.

ELIGIBILITY:
Inclusion criteria

* Adults, age > 18 years
* Spine problem for > 6 weeks, needing interdisciplinary care (risk factors, failure of first line treatment, etc)
* Inclusion in Revita program
* Informed consent to participate

Exclusion criteria

* Patients without sufficient understanding of the Dutch language
* Unable to participate in 2h rehabilitation sessions with exercises

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic spine problems in which a multidisciplinary approach is needed
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in Oswestry Disability Index (ODI) | baseline - 6 months - 1 year
  Change in functional impairment (before vs. after rehabilitation program)
  minimum score: 0 maximum score: 100 a higher score corresponds with more functional impairment
Change in pain | baseline - 6 months - 1 year
  Change in numeric rating scale (NRS) for low back/leg pain (before vs. after rehabilitation program)
  minimum score: 0 maximum score: 10 a higher score corresponds with more pain

SECONDARY OUTCOMES:
Effect on quality of life | baseline - 6 months - 1 year
  Change in EuroQoL 5D (before vs. after rehabilitation program)
  5 items with 3 levels Scale to assess health: 0-100 a higher score corresponds with better health
Effect on risk stratification tool | baseline - 6 months - 1 year
  Change in Örebro score (before vs. after rehabilitation program)
  minimum score: 0 maximum score: 100 a higher score corresponds with a higher risk profile
Effect on anxiety and depression | baseline - 6 months - 1 year
  Change in Hospital Anxiety and Depression Scale (HADS) (before vs. after rehabilitation program)
  minimum score: 0 maximum score: 21 (anxiety) - 21 (depression) a higher score corresponds with a higher suspicion for anxiety/depression
Effect on kinesiophobia | baseline - 6 months - 1 year
  Change in Tampa scale for Kinesiophobia (TSK) score (before vs. after rehabilitation program)
  minimum score: 17 maximum score: 68 a higher score corresponds with an increasing degree of kinesiophobia
Effect on fear-avoidance beliefs | baseline - 6 months - 1 year
  Change in Fear Avoidance Beliefs Questionnaire (FABQ) score (before vs. after rehabilitation program)
  minimum score: 0 maximum score: 96 a higher score corresponds with stronger fear avoidance beliefs
Effect on body awareness | baseline - 6 months - 1 year
  Change in Fremantle Back Awareness Scale Questionnaire score (before vs. after rehabilitation program)
  minimum score: 0 maximum score: 36 a higher score corresponds with a worse back-specific body perception
Treatment experience | 6 months - 1 year
  Patient Global impression of change (PGIC)
  minimum score: 1 maximum score: 7 a higher score corresponds with less impression of change
Return to Work self-efficacy | baseline - 6 months - 1 year
  "the Return to Work Self-Efficacy" questionnaire
  minimum score: 1 maximum score: 6 a higher score corresponds with a higher level of self-efficacy
Return to work | baseline - 6 months - 1 year
  number of days to return to work
Effect on functioning | baseline - 6 months - 1 year
  Change in Patient Specific Functional scale (PSFS)
  minimum score: 0 maximum score: 10 a higher score corresponds with a better functional level
Effect on medication use | baseline - 6 months - 1 year
  Change in Medication Quantification Scale (MQS)
  a higher score corresponds with a higher medication use

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: No